CLINICAL TRIAL: NCT03507829
Title: Insulin Therapy for the Prevention of New Onset Diabetes After Transplantation (ITP-NODAT) Prospective Study in Non-Diabetic De Novo Kidney Transplant Recipients
Brief Title: Insulin Therapy for the Prevention of New Onset Diabetes After Transplantation Prospective Study in Non-Diabetic De Novo Kidney Transplant Recipients
Acronym: ITP-NODAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Charite University, Berlin, Germany (Other); Medical University of Graz (Other); Hospital del Mar (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Ass.Professor Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT-Nr. 2012-000225-51
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Isophane Insulin, Human; Standard of Care; Insulin Lispro

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basal insulin (Active Comparator): NPH Insulin Titration Regimen : Pre-dinner Capillary blood glucose NPH dose initiation (IU/day) NPH dose adjustment(IU/day) > 240 mg/dl 14 Increase by 4 > 180 mg/dl 12 Increase by 4 > 140 mg/dl 10 Increase by 4 > 120 mg/dl 0 Increase by 2 100 to 119 mg/dl 0 Maintain the dose 80 - <100 mg/dl 0 Decrease by 4 60 - <80 mg/dl 0 Decrease by 8 < 60 mg/dl 0 Give ½ of previous dose
  Interventions: Drug: Human insulin isophane, Humulin N (Eli Lilly)
- Standard of care (Active Comparator): Patients assigned in this arm will receive standard of care following their kidney transplantation
  Interventions: Drug: Standard of care
- Sensor-augmented Insulin Pump (Active Comparator): Continuous subcutaneous sensor-augmented insulin-pump therapy (SAPT) with an insulin pump from Medtronic (Paradigm® Velo) for a period of approximately 3 months post-transplantation.
  Interventions: Drug: Insulin lispro, Humalog (Eli Lilly) in insulin pump

INTERVENTIONS:
Drug: Human insulin isophane, Humulin N (Eli Lilly) — Human insulin isophane, Humulin N (Eli Lilly)
  Arms: Basal insulin
Drug: Standard of care — Sliding scale short acting insulin for hyperglycemia; Sulphonylurea for NODAT
  Arms: Standard of care
Drug: Insulin lispro, Humalog (Eli Lilly) in insulin pump — Insulin lispro, Humalog (Eli Lilly) in insulin pump
  Arms: Sensor-augmented Insulin Pump

SUMMARY:
This study aims to assess the effects of early basal insulin therapy in previously non-diabetic de novo kidney transplant patients in reducing the incidence of new onset diabetes in particular and abnormal glucose metabolism in general during subsequent follow-up.The ITP NODAT study should be seen in connection with the Vienna SAPT-NODAT study (clinicaltrials.gov record number: NCT01680185), as for the final analysis, the data yielded from the three arms in those two studies will be used for an pooled analysis.

DETAILED DESCRIPTION:
New-onset diabetes after transplantation (NODAT) is strongly associated with postoperative hyperglycemia, and reduced patient as well as graft survival. In our recent proof-of-concept clinical trial (TIP), we have shown that immediate post-transplant basal insulin therapy decreases hyperglycemia and reduces the prevalence of NODAT by improving pancreatic β-cell function.

In consequence, this study as an interventional trial comparing aggressive glycemic control with early institution of insulin therapy to standard of care (dietary precaution, life-style modification, oral hypoglycemic agents and/or insulin as needed) aims to assess the effects of early basal insulin therapy in previously non-diabetic de novo kidney transplant patients in reducing the incidence of new onset diabetes in particular and abnormal glucose metabolism in general during subsequent follow-up.

Patients will be enrolled through the University of Michigan and the Medical University of Vienna, Austria (MUV), who is the official sponsor of the European part of the ITP-NODAT study. This record only refers to the European part of the ITP-NODAT study, specifically to all study patients from the following study Centers: MUV; Medical University of Graz, Austria; Charité Berlin, Germany; Hospital Del Mar, Barcelona, Spain. For the patients enrolled through the University of Michigan (i.e., the US-part of the ITP-NODAT study), a separate records exists (responsible PI: Dr. Akinlolu Ojo).

This study will involve previously non-diabetic ESRD patients undergoing kidney transplantation with either a deceased or living donor kidney who will receive standard triple immunosuppression regimen including a calcineurin inhibitor (once-daily tacrolimus in Europe, twice-daily tacrolimus in the U.S.), an anti-metabolite (mycophenolate mofetil) and corticosteroids (prednisone) and be followed at each transplant center's outpatient clinic for at least 2 years following transplantation according to the established standard center protocol.

Methods: Combining the study presented here (ITP-NODAT) and the SAPT-NODAT study mentioned above will yield three study arms, with 28 patients in each arm, namely: [1] the control arm, treated by standard-of-care; [2] the basal insulin arm, treated predominantly with intermediate acting NPH insulin (human insulin isophane, Humulin N, Eli Lilly); [3] the SAPT arm, treated with short acting insulin (Insulin lispro, Humalog, Eli Lilly), applied continuously by SAPT technology. Adult patients with absence of diabetes will be randomized prior to renal transplantation and stratified by deceased donor or living donor, if they are capable of understanding the study and are willing to give informed written consent for all three study arms. Patients will receive standard triple immunosuppressive medications (twice-daily tacrolimus, mycophenolate mofetil or mycophenolic sodium and steroids) with predefined tacrolimus targets and steroid doses. The algorithm for insulin administration is designed to account for the prominent evening peak of hyperglycemia observed in our previous TIP-study. The primary endpoint is HbA1c (in rel.%), at 3 months, and superiority will be assumed if a statistically significant difference between the SAPT-treatment group versus the standard-of-care control group can be determined, by two-sided Student's t-test. Secondary endpoints will be compared between all three groups and will include hypoglycemic events, glycemic variability, 2h glucose ≥200 mg/dL (by oral glucose tolerance test [OGTT] to determine prevalence of diabetes, prediabetes and normal glucose tolerance), beta cell function and insulin sensitivity derived from OGTT, serum creatinine, quality of life measures, patient and graft survival. All secondary endpoint comparisons relying on OGTTs will be made at 6, 12 and 24 months after kidney transplantation, respectively. The result of the 6-months OGTT will be blinded to patients and investigators to prevent subsequent treatment bias.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with end stage renal disease undergoing kidney transplantation with a deceased or living donor kidney.
2. Absence of diabetes prior to kidney transplantation, defined according to American Diabetes Association guideline (not on oral hypoglycemic agents or insulin with fasting glucose < 126 mg/dl).
3. Receiving standard triple immunosuppressive medications that include tacrolimus (once-daily in Europe, twice-daily in the U.S.), mycophenolate mofetil or mycophenolic sodium and steroids.
4. Capable of understanding the study and willing to give informed written consent for study participation.

Exclusion Criteria:

1. Patients with a diagnosis of diabetes mellitus prior to kidney transplantation, or receiving anti-diabetic medications, or having pre-transplant fasting glucose level equal or greater than 126 mg/dl on two occasions at least three days apart.
2. Patients receiving an organ transplant other than kidney.
3. Patients receiving an unlicensed drug or therapy within one month prior to study entry.
4. Patients with history of hypersensitivity to injectable insulin.
5. Patients with documented HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
incidence of NODAT | month 12 after kidney transplantation
  The incidence of NODAT 12 months after kidney transplantation defined according to American Diabetes Association criteria

SECONDARY OUTCOMES:
The incidence of NODAT at 24 months after kidney transplantation | month 24
  The incidence of NODAT at 24 months after kidney transplantation
Glycemia profile during the time of insulin therapy in arm A (intervention) comparing that of arm B (control). | week 0 to week 6
  Glycemia profile during the time of insulin therapy in arm A (intervention) comparing that of arm B (control).
The glycemia control using A1c levels, overall and among patients with NODAT, through study period 6, 12 and 24 months after kidney transplantation. | month 6, month 12, month 24
  The glycemia control using A1c levels, overall and among patients with NODAT, through study period 6, 12 and 24 months after kidney transplantation.
Incidence of impaired fasting glycemia and impaired glucose tolerance 6, 12 and 24 months after transplantation. | month 6, month 12, month 24
  Incidence of impaired fasting glycemia and impaired glucose tolerance 6, 12 and 24 months after transplantation.
Pancreatic beta-cell function at 6, 12 and 24 months after kidney transplantation, measured as insulin secretion during an OGTT in relation to the glucose stimulation (insulinogenic index - total and early phase) | month 6, month 12, month 24
  Pancreatic beta-cell function at 6, 12 and 24 months after kidney transplantation, measured as insulin secretion during an OGTT in relation to the glucose stimulation (insulinogenic index - total and early phase)
Fasting insulin resistance (mostly liver) at 6, 12 and 24 months after kidney transplantation, measured by HOMA-R and by QUICKI (insulin sensitivity) from fasting (basal) glucose and insulin concentration | month 6, month 12, month 24
  Fasting insulin resistance (mostly liver) at 6, 12 and 24 months after kidney transplantation, measured by HOMA-R and by QUICKI (insulin sensitivity) from fasting (basal) glucose and insulin concentration
Dynamic insulin sensitivity (mostly muscle and adipose tissues) at 6, 12 and 24 months after kidney transplantation, measured by OGIS and ISIcomp from OGTT data | month 6, month 12, month 24
  Dynamic insulin sensitivity (mostly muscle and adipose tissues) at 6, 12 and 24 months after kidney transplantation, measured by OGIS and ISIcomp from OGTT data
Renal function at 6, 12 and 24 months after kidney transplantation, measured by serum creatinine | month 6, month 12, month 24
  Renal function at 6, 12 and 24 months after kidney transplantation, measured by serum creatinine
Patient and graft survival 6, 12 and 24 months after kidney transplantation | month 6, month 12, month 24
  Patient and graft survival 6, 12 and 24 months after kidney transplantation
Mental component summary (MCS) and physical component summary (PCS) derived from the Kidney Disease Quality of Life Short Form (KDQoL-SFTM) at 6, 12 and 24 months after kidney transplantation | month 6, month 12, month 24
  Mental component summary (MCS) and physical component summary (PCS) derived from the Kidney Disease Quality of Life Short Form (KDQoL-SFTM) at 6, 12 and 24 months after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, MD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwaiger E, Krenn S, Kurnikowski A, Bergfeld L, Perez-Saez MJ, Frey A, Topitz D, Bergmann M, Hodlmoser S, Bachmann F, Halleck F, Kron S, Hafner-Giessauf H, Eller K, Rosenkranz AR, Crespo M, Faura A, Tura A, Song PXK, Port FK, Pascual J, Budde K, Ristl R, Werzowa J, Hecking M. Early Postoperative Basal Insulin Therapy versus Standard of Care for the Prevention of Diabetes Mellitus after Kidney Transplantation: A Multicenter Randomized Trial. J Am Soc Nephrol. 2021 Aug;32(8):2083-2098. doi: 10.1681/ASN.2021010127. PMID 34330770